CLINICAL TRIAL: NCT06519838
Title: Effect of Pre-Warming of Local Anesthesia in Reducing Pain Perception During Injection in Children: A Randomized Controlled Clinical Trial
Brief Title: Effect of Pre-Warming of Local Anesthesia in Reducing Pain Perception During Injection in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Emad (Other)
Responsible Party: Sponsor-Investigator, Andrew Emad, Pediatric Dentist, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1/2023
Record Dates: First submitted 2024-07-14; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Local Anesthesia; Dental Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Maxillary infiltration at room temperature (Active Comparator)
  Interventions: Other: Local anesthesia solution at room temperature; Other: Maxillary infiltration technique
- Inferior alveolar nerve block at room temperature (Active Comparator)
  Interventions: Other: Local anesthesia solution at room temperature; Other: Inferior alveolar nerve block technique
- Maxillary infiltration pre-warmed to 37°C (Experimental)
  Interventions: Other: Local anesthesia solution pre-warmed to 37°C; Other: Maxillary infiltration technique
- Inferior alveolar nerve block pre-warmed to 37°C (Experimental)
  Interventions: Other: Local anesthesia solution pre-warmed to 37°C; Other: Inferior alveolar nerve block technique
- Maxillary infiltration pre-warmed to 40°C (Experimental)
  Interventions: Other: Local anesthesia solution pre-warmed to 40°C; Other: Maxillary infiltration technique
- Inferior alveolar nerve block pre-warmed to 40°C (Experimental)
  Interventions: Other: Local anesthesia solution pre-warmed to 40°C; Other: Inferior alveolar nerve block technique

INTERVENTIONS:
Other: Local anesthesia solution at room temperature — The local anesthesia cartridge is used at room temperature (average of 21 °C)
  Arms: Inferior alveolar nerve block at room temperature; Maxillary infiltration at room temperature
Other: Local anesthesia solution pre-warmed to 37°C — About 150 ml of water at 21°C is added to the heating compartment of the heating device. The Local anesthesia cartridge is placed at the bottom of the heating compartment. The device is plugged in and the control gauge is set at the "Express milk warming setting for contents up to 180ml/6oz" mark. The contents would reach 37°C at 120 seconds.
  Arms: Inferior alveolar nerve block pre-warmed to 37°C; Maxillary infiltration pre-warmed to 37°C
Other: Local anesthesia solution pre-warmed to 40°C — About 150 ml of water at 21°C is added to the heating compartment of the heating device. The Local anesthesia cartridge is placed at the bottom of the heating compartment. The device is plugged in and the control gauge is set at the "Express milk warming setting for contents up to 180ml/6oz" mark. The contents would reach 40°C at 130 seconds.
  Arms: Inferior alveolar nerve block pre-warmed to 40°C; Maxillary infiltration pre-warmed to 40°C
Other: Maxillary infiltration technique — A 30 gauge short needle is oriented so that the bevel is facing the bone. The syringe is held parallel to the long axis of the tooth and the needle is inserted into the height of the mucobuccal fold over the offending tooth. The needle is advanced to a depth of 1 millimeter into the tissues. Aspiration is done, and once it is negative then 0.6 ml (nearly one third of the cartridge) of the anesthetic solution is injected slowly without permitting the tissues to balloon.
  Arms: Maxillary infiltration at room temperature; Maxillary infiltration pre-warmed to 37°C; Maxillary infiltration pre-warmed to 40°C
Other: Inferior alveolar nerve block technique — While the mouth is opened as wide as possible, the index finger palpates the external oblique ridge reaching the Coronoid notch. A 27-gauge long dental needle will be used for injection. The needle will be directed between the two primary molars on the opposing side of the arch, penetrating the tissues at the point halfway between coronoid notch and the pterygomandibular raphe at the occlusal plane level or slightly lower.The needle is withdrawn 2mm to aspirate. Once negative aspiration is checked, the remainder of the solution is deposited slowly. Approximately 1.0 mL of LA will be delivered near the inferior alveolar nerve. The average depth of insertion is about 15mm, which is nearly two-thirds the needle length.
  Arms: Inferior alveolar nerve block at room temperature; Inferior alveolar nerve block pre-warmed to 37°C; Inferior alveolar nerve block pre-warmed to 40°C

SUMMARY:
The aim of the current study was to evaluate the pain perception upon injection of pre-warmed dental anesthetic solution (at 370C and 400C) versus that at room temperature (Average 23 degrees) during Maxillary Infiltration and Mandibular Inferior Alveolar Nerve Block techniques in children

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients with ASA 1 or 2 Classification.
* Patients with Frankl Behavior Classification 3-4.
* Patients having at least one carious primary molar that requires dental treatment under the effect of local anesthesia.
* Parents' willingness to participate through informed written consent.

Exclusion Criteria:

* Patients with previous negative dental experience.
* Patients complaining of cellulitis or infection spreading in the fascial spaces.
* Patients who have received analgesics within the previous 12 hours before receiving the required dental treatment.
* Patients with any Intellectual Impairment.
* Patients with a history of allergy from any of the components of the dental anesthetic carpule.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Heart rate (HR) monitoring | during local anesthesia administration
  A pulse oximeter will be used to record and measure the patient's heart rate. A baseline reading will be obtained before the LA administration and another reading will be obtained directly after the injection is carried out. Heart rate ranging between 70-100 is considered normal.
Pain during injection using Sound, Eye, Motor (SEM) Scale | during local anesthesia administration
  Sound, Eye, Motor (SEM) Scale was used as an objective mean to assess pain during local anesthesia administration. It comprises the following parameters:
  * Sound
  * Eye
  * Bodily movements The slightest changes in the sound, eye movement and bodily movement of the patient will be categorized as one of the following levels; comfortable, mild, moderate, and severe discomfort and hence given a grade of 1, 2, 3 or 4 respectively. The final SEM score will be calculated by adding the grades of the three parameters.
Pain during injection using Face scale | during local anesthesia administration
  To assess pain subjectively during local anesthesia administration, a modified face scale. It consists of three schematic faces with different facial expressions for happy and sad faces representing:
  1. Satisfaction
  2. Indifference
  3. Dissatisfaction Each patient was trained on using the scale by modelling and then requesting from every patient to think of the last time she/he went through a painful experience and to choose the facial expression that best relates his/her current experience of discomfort to the previous one

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt